CLINICAL TRIAL: NCT04499404
Title: A WeChat-based Intervention to Promote and Support Breastfeeding in China: A Multi-center Randomized Controlled Trial
Brief Title: A WeChat-based Intervention to Support Breastfeeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chengdu Jinjiang Maternity and Child Health Hospital (Other)
Collaborators: Chengdu Women's and Children's Central Hospital (Other); Curtin University (Other)
Responsible Party: Principal Investigator, Li Tang, Assistant Professor, Chengdu Jinjiang Maternity and Child Health Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2019FYH014
Record Dates: First submitted 2020-07-28; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Exclusive Breastfeeding
Keywords: exclusive breastfeeding; complementary feeds; smart phone application; randomized controlled trial; WeChat
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants receive breastfeeding-related information from WeChat
  Interventions: Other: Breastfeeding related information delivered by WeChat
- Control group (Active Comparator): Participants receive non-breastfeeding information from WeChat
  Interventions: Other: Non-breastfeeding related information delivered by WeChat

INTERVENTIONS:
Other: Breastfeeding related information delivered by WeChat — Participants in the intervention group will be asked to follow our WeChat public account immoderately after randomization. They will receive breastfeeding related messages three times a week from WeChat, including preparation for breastfeeding after birth and the health benefits of breastfeeding, from baseline until childbirth. After childbirth, intervention group mothers will continue to receive information, which is mainly about breastfeeding, once a week for 6 months. WeChat will send push notifications to remind mothers about the importance of exclusive breastfeeding, build confidence and motivate them to continue exclusive breastfeeding.
  Arms: Intervention group
Other: Non-breastfeeding related information delivered by WeChat — Participants in the control group will be asked to follow our WeChat public account immoderately after randomization. They will receive messages mainly on topics of healthy lifestyle and nutrition during pregnancy, from baseline until childbirth. After childbirth, they will continue to receive information on other topics of interest to mothers, such as immunization, safety, infant growth, and etc., until 6 months postpartum.
  Arms: Control group

SUMMARY:
The aim of the randomized controlled trial (RCT) is to evaluate the effects of an intervention program delivered via WeChat platform to support exclusive breastfeeding in China. WeChat, a free smart phone application, is the most popular social networking platform in China. It will be used to deliver health educational messages to the study participants. Our hypothesis is that the intervention program can lead to at least a 10% increase in exclusive breastfeeding prevalence at 6 months when compared to the control group.

A multicenter RCT of 1,000 participants will be conducted at four maternity hospitals in Chengdu, China. Eligible pregnant women who consent to participate will be recruited from the antenatal clinic at around 30 weeks of gestation and will be randomly assigned to either the intervention or control group on a 1:1 ratio.

After randomization, all participants will be asked to scan a Quick Response code to follow our WeChat public account, which can send push notifications to alert participants for new content, topics, links to a searchable library and frequently asked questions and answers. From baseline until childbirth, control group participants will receive non-breastfeeding related messages, such as healthy lifestyle and nutrition during pregnancy, from WeChat, whereas the intervention group participants will receive breastfeeding related messages, including preparation for breastfeeding after birth and the health benefits of breastfeeding, from WeChat. After childbirth, intervention group mothers will continue to receive information about breastfeeding for 6 months. The investigators will use WeChat to remind mothers about the importance of exclusive breastfeeding, build confidence and motivate them to continue exclusive breastfeeding. Meanwhile, the control group participants will receive information on other topics of interest to mothers, such as immunization, safety, infant growth, and etc.

Each participant will be interviewed in person by trained nurses at baseline, at discharge and be interviewed by telephone using structured questionnaires at 1, 4, and 6 months postpartum to collect detailed information on breastfeeding practices. All participants receive normal prenatal and postpartum maternity services. Cox proportional hazard models and multilevel mixed regression models will be performed respectively to compare the duration of exclusive breastfeeding and the rates of exclusive breastfeeding within six months postpartum between intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* own a smart phone;
* 18 years or above;
* sufficient language skills (completed secondary school education);
* carry a singleton fetus;
* at a gestational age of 28 to 30 weeks;

Exclusion Criteria:

* have existing medical conditions or pregnancy complications which may inhibit breastfeeding initiation, according to their medical doctor;
* intend to give birth in health institutes other than the study hospitals.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-06-28 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Exclusive breastfeeding rate at 6 months postpartum | 6 months postpartum
  Breastfeeding while giving no other food or liquid, not even water, with the exception of drops or syrups consisting of vitamins, mineral supplements or medicines.
Full breastfeeding rate at 6 months postpartum | 6 months postpartum
  Infants who are receiving almost all of their nutrients from breast milk but take some other liquids such as water, water-based drinks, oral rehydration solutions, ritual fluids, and drops or syrups.

SECONDARY OUTCOMES:
Infant's first feed | 0-7 days postpartum
  % of infants fed with breastmilk as their first feed
Exclusive breastfeeding duration to 4 months postpartum | 0-4 months postpartum
  Breastfeeding while giving no other food or liquid, not even water, with the exception of drops or syrups consisting of vitamins, mineral supplements or medicines.
Exclusive breastfeeding duration to 6 months postpartum | 0-6 months postpartum
  Breastfeeding while giving no other food or liquid, not even water, with the exception of drops or syrups consisting of vitamins, mineral supplements or medicines.
Rate of early introduction of complementary feeding | 0-4 months postpartum
  Complementary feeding is defined as feeding infants with solid foods and liquids other than breastmilk or infant formula.
Any breastfeeding duration to 6 months postpartum | 0-6 months postpartum
  The child has received breastmilk (direct from the breast or expressed) with or without other drink, formula or other infant food

CONTACTS AND LOCATIONS:
Overall Officials: Li Tang, PhD, Principal Investigator — Chengdu Jinjiang Maternity and Child Health Hospital
Locations (1):
- Chengdu Qingyang Maternal and Child Health Hospital, Chengdu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tang L, Lee AH, Binns CW, Duan L, Liu Y, Li C. WeChat-based intervention to support breastfeeding for Chinese mothers: protocol of a randomised controlled trial. BMC Med Inform Decis Mak. 2020 Nov 19;20(1):300. doi: 10.1186/s12911-020-01322-8. PMID 33213446